CLINICAL TRIAL: NCT00544817
Title: A Phase II Trial of Concurrent Radiation Therapy and Temozolomide Followed by Temozolomide Plus Sorafenib in the First-Line Treatment of Patients With Glioblastoma Multiforme
Brief Title: Radiation Therapy and Temozolomide Followed by Temozolomide Plus Sorafenib for Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CNS 09
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Glioblastoma Multiforme
Keywords: Concurrent Radiation Therapy; Temozolomide; Sorafenib; First-line; Glioblastoma Multiforme; Phase II
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy (Experimental): In the combined modality portion of the study, patients were administered:
  Radiation Therapy - 2 Gy/fraction, Single daily fractions M-F, to 60 Gy total Temozolomide - 75 mg/m2 by mouth once daily
  Patients took a four week break before beginning follow-up systemic therapy:
  Temozolomide - 150 mg /m2 by mouth on days 1-5 every 28 days for 6 cycles Sorafenib - 400 mg by mouth twice a day for 6 months
  Interventions: Radiation: Radiation Therapy; Drug: Temozolomide; Drug: Sorafenib

INTERVENTIONS:
Radiation: Radiation Therapy — 2 Gy/fraction, single daily fractions M-F, to 60 Gy total
Drug: Temozolomide — In Combined Modality Therapy, administered as 75 mg/m2 by mouth once daily
  In follow-up systemic therapy, administered as 150 mg/m2 by mouth on days 1-5 every 28 days for 6 cycles
  Other Names: Temodar
Drug: Sorafenib — In follow-up systemic therapy, administered as 400 mg by mouth twice daily for 6 months
  Other Names: Nexavar

SUMMARY:
The mechanism of action of sorafenib makes it an interesting drug to investigate in the treatment of patients with glioblastoma multiforme. Efficacy of agents with anti-angiogenic activity has already been demonstrated and the PDGF receptor target may also be pertinent in glioblastoma. The combination of temozolomide plus sorafenib has been investigated previously in the treatment of patients with advanced melanoma. The combination was generally well tolerated; in previously untreated patients, a standard dose of sorafenib (400mg PO bid) was administered with temozolomide 150mg/m2 PO daily for 5 days, repeated every 28 days (23).

In this multicenter phase II study, patients with newly diagnosed glioblastoma will receive standard treatment, including initial debulking surgical resection (if feasible) followed by high-dose radiation therapy with concurrent temozolomide. After completion of radiation therapy, patients will continue treatment with temozolomide (150mg/m2 days 1-5) and sorafenib (400mg PO bid daily), repeated at 28-day intervals for 6 cycles.

DETAILED DESCRIPTION:
All patients entering this study will initially undergo combined modality treatment with concurrent radiation therapy + temozolomide. Four weeks after completing radiation therapy, patients will begin 6 months of follow-up treatment with oral temozolomide plus sorafenib.

Combined Modality Therapy - Radiation Therapy Radiotherapy must begin within ≤ 6 weeks of surgery. One treatment of 2.0Gy will be given daily 5 days per week for a total of 60.0Gy over 6 weeks. Temozolomide 75mg/m2 PO will be given daily, beginning on the first day of radiation therapy and continuing through the last day of radiation therapy.

After completion of combined modality therapy, patients will have 4 weeks without any therapy.

Systemic Therapy Beginning 4 weeks after the completion of radiation therapy, patients will receive 6 months of treatment with temozolomide and sorafenib. Temozolomide 150mg/m2 orally will be administered days 1-5, and repeated every 28 days for 6 courses. Sorafenib 400mg PO bid will be administered on days 1-28, repeated for 6 courses concurrently with temozolomide

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed intracranial glioblastoma multiforme (WHO grade 4).
2. Patients who have had partial or complete surgical debulking are eligible, as are those with inoperable glioblastoma.
3. No previous treatment for glioblastoma except for previous surgical debulking (i.e. no previous radiotherapy, local chemotherapy, or systemic therapy).
4. ECOG performance status 0 or 1 (See Appendix C)
5. Age ≥ 18 years
6. Adequate bone marrow function: hemoglobin ≥ 9.0g/dL; ANC ≥ 1500/μL; platelet count ≥ 100,000/μL.
7. Adequate liver function

   * Total bilirubin ≤ 1.5 x ULN
   * ALT and AST ≤ 2.5 x ULN
8. Serum creatinine < 1.5 x ULN
9. Women of child-bearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Women must agree to not breast feed while receiving study treatment.
10. Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control) while receiving study treatment. Women should use adequate birth control for at least 3 months after the last administration of sorafenib.
11. INR < 1.5 or PT/PTT within normal limits in patients not receiving anticoagulation. However, patients receiving anticoagulation treatment with an agent such as warfarin or heparin are also eligible. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
12. Patients must have the ability to understand and the willingness to sign written informed consent. A signed informed consent must be obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Patients must have the ability to swallow whole pills.
2. Active cardiac disease: congestive heart failure > class 2 NYHA (Appendix D); unstable angina or new onset angina within the last 3 months; myocardial infarction within the last 6 months.
3. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
4. Uncontrolled hypertension defined as systolic blood pressure > 150mm Hg or diastolic pressure > 90mm Hg, despite optimal medical management
5. Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C infection
6. Active clinically serious infection > grade 2
7. Thrombotic or embolic events including cerebral vascular accident or TIAs within the past 6 months
8. Pulmonary hemorrhage/bleeding event ≥ grade 2 within 4 weeks of the first dose of sorafenib
9. Any other hemorrhage/bleeding event ≥ grade 3 within 4 weeks of the first dose of sorafenib
10. Serious non-healing wound, ulcer, or bone fracture
11. Evidence or history of bleeding diathesis or coagulopathy
12. Major surgery, open biopsy, or significant traumatic injury within 4 weeks of beginning treatment with sorafenib
13. Use of St. John's Wort or rifampicin
14. Known or suspected allergy to sorafenib or temozolomide
15. Any malabsorption problem
16. Other active malignancies, or treatment for invasive cancer within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Result] Hainsworth JD, Ervin T, Friedman E, Priego V, Murphy PB, Clark BL, Lamar RE. Concurrent radiotherapy and temozolomide followed by temozolomide and sorafenib in the first-line treatment of patients with glioblastoma multiforme. Cancer. 2010 Aug 1;116(15):3663-9. doi: 10.1002/cncr.25275. PMID 20564147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2007 and July 2008, 47 patients were enrolled
Period: Combined Modality
Arm/Group | Combination Therapy
Started | 47
Completed | 40
Not Completed | 7
Not completed — Lack of Efficacy | 2
Not completed — Worsening Neurologic Symptoms | 2
Not completed — Adverse Event | 2
Not completed — Intercurrent Illness - Pneumonia | 1
Period: No Treatment Interval
Arm/Group | Combination Therapy
Started | 40
Completed | 28
Not Completed | 12
Not completed — Lack of Efficacy | 8
Not completed — Physician Decision | 3
Not completed — Adverse Event | 1
Period: Follow-up Systemic Therapy
Arm/Group | Combination Therapy
Started | 28
Completed | 9
Not Completed | 19
Not completed — Lack of Efficacy | 15
Not completed — Physician Decision | 3
Not completed — Intercurrent Illness - Pneumonia | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 47
Months | 6 [3.7 to 7]

2. Secondary Outcome: Overall Survival
Description: Defined as Day 1 of protocol treatment to date of death from any cause.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 47
Months | 12 [7.2 to 16]

3. Secondary Outcome: Objective Response
Description: The number of patients with complete or partial responses measured from the time of initial response to documented tumor progression. Radiologic response was defined using the Macdonald criteria.
  The Macdonald criteria divides response into 4 types of response based on imaging (MRI) and clinical features, as follows: 1) complete response (CR); 2) partial response (PR); 3) stable disease (SD); and 4) progression (PD).
  Criteria:
  CR: disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks, no new lesions. No corticosteroids, clinically stable or improved.
  PR: >=50% decrease of all measurable enhancing lesions, sustained for at least 4 weeks, no new lesions. Stable or reduced corticosteroids, clinically stable or improved.
  SD: does not qualify for complete response, partial response or progression. Clinically stable.
  PD: >= 25% increase in enhancing lesions, any new lesions. Clinical deterioration.
Time Frame: every 8 weeks until disease progression, estimated 18 months
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 47
participants | 13

ADVERSE EVENTS:
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 19/47
Other Adverse Events (participants affected / at risk) | 32/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=47)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Acute radiation encephalopathy (Nervous system disorders) | 1 (1)
Dilantin toxicity (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Seizure (Nervous system disorders) | 2 (2)
Decreased LOC (Nervous system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
DVT (Vascular disorders) | 1 (1)
INR (Blood and lymphatic system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Steroid-induced weakness (General disorders) | 1 (1)
Mental status changes (Nervous system disorders) | 1 (1)
Speech impairment (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral pulmonary emboli (Vascular disorders) | 1 (1)
Septicemia (Infections and infestations) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=47)
Rash - Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 10 (17)
Fatigue (General disorders) | 32 (63)
Rash (Skin and subcutaneous tissue disorders) | 20 (35)
Nausea (Gastrointestinal disorders) | 21 (35)
Diarrhea (Gastrointestinal disorders) | 11 (15)
Vomiting (Gastrointestinal disorders) | 10 (13)
Hypertension (Cardiac disorders) | 4 (5)
Hair loss/Alopecia (Skin and subcutaneous tissue disorders) | 20 (37)
ALT/SGPT (Metabolism and nutrition disorders) | 4 (8)
Anorexia (Gastrointestinal disorders) | 18 (30)
Bicarbonate serum-low (Metabolism and nutrition disorders) | 3 (3)
Vision - Blurred Vision (Eye disorders) | 5 (5)
Confusion (Nervous system disorders) | 17 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (4)
Taste Alteration (dysgeusia) (Gastrointestinal disorders) | 6 (10)
Dysphagia (Gastrointestinal disorders) | 3 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema: Head and Neck (Blood and lymphatic system disorders) | 3 (4) — Face
Edema: Limb (Blood and lymphatic system disorders) | 7 (12)
Fever (General disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 11 (15)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (5)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (13)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (6)
Metablolic/Laboratory - Other (hypobilirubinemia) (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (4)
Incontinence, urinary (Renal and urinary disorders) | 3 (3)
Infection - Other, Lung (pneumonia) (Infections and infestations) | 3 (4)
Infection - Other, Urinary Tract NOS (Renal and urinary disorders) | 4 (6)
Insomnia (General disorders) | 7 (14)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 13 (24)
Memory Impairment (Nervous system disorders) | 4 (7)
Mood Alteration, Anxiety (Nervous system disorders) | 7 (9)
Mood Alteration, Depression (Nervous system disorders) | 7 (9)
Mucositis (Gastrointestinal disorders) | 3 (5)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 12 (17)
Seizure (Nervous system disorders) | 11 (12)
Neuropathy: Motor (Nervous system disorders) | 9 (19)
Neuropathy: Sensory (Nervous system disorders) | 3 (9)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 (6)
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 (3)
Pain - Headache (Nervous system disorders) | 18 (24)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain - Pain NOS (General disorders) | 8 (11)
Personality/behavioral (Nervous system disorders) | 5 (5)
Platelets (Blood and lymphatic system disorders) | 16 (28)
Somnolence/depressed level of consciousness (Nervous system disorders) | 6 (7)
Speech Impairment (Nervous system disorders) | 11 (18)
Tremor (Nervous system disorders) | 4 (4)
Weight Loss (General disorders) | 5 (11)
Constipation (Gastrointestinal disorders) | 10 (17)
Erythema (Musculoskeletal and connective tissue disorders) | 3 (7)
Infection - Thrush (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.